CLINICAL TRIAL: NCT01024257
Title: Pterygium Treatment Using Single Beta-therapy as Adjuvant Treatment Compared to Conjunctival Autograft
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Marilia Medicine School (Other)
Other Study IDs: Famema0010
Record Dates: First submitted 2009-11-30; First posted 2009-12-02 (Estimated); Last update posted 2009-12-02 (Estimated); Status verified 2009-12

CONDITIONS: Pterygium
Keywords: beta-irradiation;conjunctival autograft;pterygium;recurrence; clinical trial
MeSH Terms: conditions — Pterygium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- conjunctival autograft plus beta-irradiation (Experimental)
  Interventions: Radiation: beta-irradiation
- conjunctival autograft (Active Comparator)
  Interventions: Procedure: conjunctival autograft

INTERVENTIONS:
Radiation: beta-irradiation
  Arms: conjunctival autograft plus beta-irradiation
Procedure: conjunctival autograft
  Arms: conjunctival autograft

SUMMARY:
PURPOSE: To affirm the effectiveness and complication rate of postoperative single-dose beta-irradiation (RT) with (90) Sr in the case of primary pterygium in a clinical trial. METHODS AND MATERIALS: This trial was designed as a prospective, randomized, single center study. Surgery was performed in all cases according to the conjunctival autograft technique. One thousand and four patients with 108 pterygia were postoperatively randomized to either beta-RT or observation. In the case of beta-RT, a (90) Sr eye applicator was used to deliver 1000 cGy to the sclera surface at a dose rate of between 200 and 250 cGy/min. After treatment, both an ophthalmologist and a radiation oncologist performed the follow-up examinations. The accumulated data were analyzed using a group sequential test. RESULTS: Between February 2007 and September 2008, 104 eyes with primary pterygium were operated on according to the trial protocol. Additional treatment was performed within 24 hours postoperatively. Four patients were lost to follow-up, resulting in 104 patients who could be analyzed. In the 54 eyes randomized to receive beta-RT, 5 relapses occurred compared with 8 recurrences in the 50 eyes that no received RT, for a crude control rate of 90.7 % vs. 84 %, respectively. At a mean follow-up of 9 months (range 4- 18), major treatment complications had not been observed . CONCLUSION: Single-dose beta-RT of 1000cGy after conjunctival autograft surgery is a simple, effective, and safe treatment that reduces the risk of primary pterygium recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Fresh pterygium without previous treatment.
* Adult patients with age higher than 18 years.

Exclusion Criteria:

* Diagnosis of glaucoma.
* Previous treatment of pterygium.
* Patients with age less than 18 years old.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Gustavo Viani Arruda, Marília, Saop Paulo, Brazil